CLINICAL TRIAL: NCT04524195
Title: A Study of PET Imaging of T-cell Activation With [18F]F-AraG in Advanced Non-small Cell Lung Cancer (NSCLC) Patients Undergoing PD-1/PD-L1-directed Therapy
Brief Title: PET Imaging With [18F]F-AraG in Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is terminated because the PI left the institution.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: CellSight Technologies, Inc. (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J19119; IRB00208724 (Other: JHM IRB)
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: J19119; PET/CT; [18F]F-AraG; NSCLC; PD-1; PD-L1; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]F-AraG (Experimental): A one-time nominal injection dose of 5 millicurie (mCi) +/- will be administered at each PET/CT imaging time point.
  Interventions: Drug: [18F]F-AraG Injection

INTERVENTIONS:
Drug: [18F]F-AraG Injection — Single dose of 5 mCi+/- [18F]F-AraG IV injection followed by the PET/CT scan. A baseline [18F]F-AraG PET/CT will be performed at about 0-7 days before patient receives the first dose of PD-1/PD-L1 immunotherapy. A second [18F]F-AraG PET-CT will be performed at less than 14 days after the first dose of PD-1/PD-L1 immunotherapy is administered and before the second dose of PD-1/PD-L1 immunotherapy is given.

SUMMARY:
This is a prospective, single center, single-arm clinical trial in 20 patients with non-small cell lung cancer (NSCLC) undergoing PD-1/PD-L1-directed therapy. This research is being done to find out if the radioactive compound called [18F]F-AraG is a helpful imaging agent for detecting changes in cancer's anti-tumor immune response (or activation of T-cell) levels for non-small cell lung cancer (NSCLC) patients who will receive a cancer immunotherapy regimen (immunotherapy works by encouraging the body's own immune system to attack the cancer cells).

DETAILED DESCRIPTION:
The purpose of this study is to find out how the radiotracer called [18F]F-AraG can help investigate changes in cancer's anti-tumor immune response (or activation of T-cell) levels during positron emission tomography (PET) scans. [18F]F-AraG has the potential to serve as a noninvasive imaging biomarker in the monitoring of T-cell mediated anti-tumor immune response following administration of an immunotherapeutic agent.

Participants in this study will have tests, exams and procedures that are for study purposes. Participants will be in this study up to one month which will include about three clinic visits.

A baseline [18F]F-AraG PET-CT will be obtained 0-7 days before a NSCLC patient receives PD-1/PD-L1 immunotherapy. A second [18F]F-AraG PET-CT will be performed 10-14 days after PD-1/PD-L1 immunotherapy is administered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and willing and able to provide informed consent.
* Subjects with stage I, II, or III A NSCLC and plan to receive neoadjuvant PD-1/PD-L1 immunotherapy with an intention for curative surgery. Subjects will be receiving neoadjuvant immunotherapy through enrollment in therapeutic clinical trials
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at the time of enrollment.
* For females of childbearing potential, negative serum pregnancy test within a 10 day period will be obtained prior to PET study.

Exclusion Criteria:

* Severe impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73 m2 and/or on dialysis.
* Pregnant female patients; breastfeeding female patients.
* Any medical condition that in the opinion of the study investigators would constitute a safety risk to the subject.
* Any investigational radiation exposure in the past calendar year that in combination with the radiation exposure from this study would exceed 5 rem.
* Administered a radioisotope ≤5 physical half-lives prior to the day of PET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Percent Change in uptake of [18F]F-AraG before and after one dose of anti-PD-L1 | Baseline and 10-14 days after first dose of neoadjuvant therapy
  Percent Change in standard uptake value (SUV) of [18F]F-AraG PET-CT imaging of primary tumor and of lymph nodes at baseline to after the first dose of neoadjuvant therapy.
Percent pathologic response at the time of surgery | At the time of surgery
  100% minus the percentage of viable tumor remaining in the tumor bed.
Correlation between [18F]F-AraG uptake and percent pathologic response as assessed by the Spearman correlation coefficient | 5 years
  Spearman correlation coefficient will be calculated in assessing the correlation between [18F]F-AraG uptake and pathologic response.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pomper, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No